CLINICAL TRIAL: NCT02177500
Title: An Eight Week Randomized, Double-Blind Study Comparing a Fixed Dose Combination of Telmisartan 40 mg Plus Hydrochlorothiazide 12.5 mg to Telmisartan 40 mg in Patients Who Fail to Respond Adequately to Treatment With Telmisartan 40 mg
Brief Title: Telmisartan Plus Hydrochlorothiazide in Subjects With Mild-to-moderate Hypertension Who Failed to Respond to Telmisartan Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.323
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan, hydrochlorothiazide drug combination; Telmisartan

ARMS (2):
- Telmisartan + hydrochlorothiazide and matching placebo (Experimental)
  Interventions: Drug: Telmisartan + hydrochlorothiazide; Drug: Placebo
- Telmisartan and matching placebo (Experimental)
  Interventions: Drug: Telmisartan; Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan + hydrochlorothiazide
  Arms: Telmisartan + hydrochlorothiazide and matching placebo
Drug: Telmisartan
  Arms: Telmisartan and matching placebo
Drug: Placebo

SUMMARY:
An eight week study to compare the effect of a fixed dose combination of Telmisartan 40 mg plus hydrochlorothiazide (HCTZ) 12.5 mg to Telmisartan 40 mg alone on diastolic and systolic blood pressure in patients who fail to respond adequately to telmisartan monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* History of mild-to-moderate hypertension
* Patients who fail to respond adequately to telmisartan monotherapy
* Participants between 18 and 80 years of age
* Willingness and ability to provide written informed consent

Exclusion Criteria:

* Patients taking more than three anti-hypertensive medications at the screening visit
* Pre-menopausal women

  * Who are not surgically sterile
  * Who are NOT practicing acceptable means of birth control or who do NOT plan to continue using an acceptable method throughout the study. Acceptable methods of birth control include intrauterine device (IUD), oral, implantable or injectable contraceptives
* Any women:

  * Who has a positive serum pregnancy test at screening (Visit 1) or baseline (Visit 3)
  * Who is nursing
* Hepatic and/or renal dysfunction as defined by the following laboratory parameters

  * SGPT (serum glutamate pyruvate transaminase) or SGOT (serum glutamate oxaloacetate transaminase) greater than two times the upper limit of normal
  * Serum creatinine > 2.3 mg/dL
* Clinically relevant sodium depletion, hyperkalemia, or hypokalemia at baseline
* Known or suspected secondary hypertension
* Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; post-renal transplant patients, presence of only one functioning kidney
* Congestive heart failure (CHF) (NYHA (New York Heart Association) functional class CHF III-IV)
* Unstable angina within the past three months
* Stroke within the past six months
* Myocardial infarction or cardiac surgery within the past three months
* PTCA (percutaneous transluminal coronary angioplasty) within the past three months
* History of symptoms characteristic of angioedema during treatment with ACE inhibitors, angiotension II antagonists, thiazide diuretics, β-blockers or calcium channel blockers
* Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator
* Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
* Administration of digoxin or other digitalis-type drugs
* Patients with Type I or Type II diabetes mellitus whose diabetes has not been stable and controlled for at least the past three months as defined by an HbA1C ≥ 10%
* Known drug or alcohol dependency within the past one year period
* Concomitant administration of medications known to affect blood pressure, except medications allowed by the protocol
* Patients receiving any investigational therapy within one month of signing the informed consent form. Patients who have participated in previous telmisartan (except if they were on the fixed dose combination in the 502.261 study or enrolled in the 502.321 open-label extension study) studies may participate in this study provided there has been at least one month between discontinuing the previous study and signing the consent for the present study
* Known hypersensitivity to any component of the formulations
* Any clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of trial medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2000-01; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in seated diastolic blood pressure (DBP) | baseline and after 8 weeks of treatment

SECONDARY OUTCOMES:
Change from baseline in seated systolic blood pressure (SBP) | baseline and after 8 weeks of treatment
Blood pressure control | 8 weeks
Systolic blood pressure response | 8 weeks
Incidence of adverse events | up to 16 weeks
Change from baseline in physical examination | Baseline and day 56
Change from baseline in heart rate | Baseline, day 28 and 56
Change from baseline in laboratory parameters | Baseline and day 56
Change from baseline in 12-lead ECG (electrocardiogram) | Baseline and day 56